CLINICAL TRIAL: NCT02543853
Title: The Effect of Two Different Endoscopic Entry Techniques on Postoperative Gastrointestinal Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, enis ozkaya, Assoc. Prof., Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 990902
Record Dates: First submitted 2015-05-24; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Gastrointestinal Disorder Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- veres needle entry arm (Active Comparator): Vere needle will be used to provide penumoperiteum than postoperative gastrointestinal functions will be compared
  Interventions: Other: veres needle entry
- direct trocar entry arm (Active Comparator): Direct trocar entry will be used to provide penumoperiteum than postoperative gastrointestinal functions will be compared
  Interventions: Other: direct trocar entry

INTERVENTIONS:
Other: direct trocar entry — direct trocar entry to provide pneumoperitoneum
  Arms: direct trocar entry arm
Other: veres needle entry — veres needle entry to provide pneumoperitoneum
  Arms: veres needle entry arm

SUMMARY:
The purpose of this study is to determine effect of veres needle entry and direct trocar entry on postoperative gastrointestinal functions.

DETAILED DESCRIPTION:
Women planned to have laparoscopic surgery will be randomized into two groups, in first group pneumoperitoneum will be provided by veres needle, in other group direct trocar entry will be used to provide pneumoperitoneum. After surgery gastrointesitinal functions, shoulder pain, blood loss will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic surgery for benign or malignant disease

Exclusion Criteria:

* Patients with gastrointestinal intervention
* Patients who had undergone previous operations
* Patients with gastrointestinal intervention dysfunction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Bowel sound (first bowel sound) | Postoperative first 72 hours
  time from surgery to first bowel sound as hours

SECONDARY OUTCOMES:
Gas discharge | Postoperative first 72 hours
  time from surgery to first bowel sound as hours

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Compeau C, McLeod NT, Ternamian A. Laparoscopic entry: a review of Canadian general surgical practice. Can J Surg. 2011 Oct;54(5):315-20. doi: 10.1503/cjs.011210. PMID 21774882
- [Background] Daskalakis M, Scheffel O, Weiner RA. High flow insufflation for the maintenance of the pneumoperitoneum during bariatric surgery. Obes Facts. 2009;2 Suppl 1(Suppl 1):37-40. doi: 10.1159/000198252. Epub 2009 Mar 18. PMID 20124777
- [Result] Ahmad G, O'Flynn H, Duffy JM, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD006583. doi: 10.1002/14651858.CD006583.pub3. PMID 22336819